CLINICAL TRIAL: NCT01295541
Title: Early Progressive Mobility in the CVICU: Assessing Current Status
Status: Completed | Type: Observational
Sponsor: Hill-Rom (Industry)
Responsible Party: Catherine VanGilder, Hill-Rom
Other Study IDs: CR-2009-05a
Record Dates: First submitted 2010-07-06; First posted 2011-02-14 (Estimated); Last update posted 2011-02-14 (Estimated); Status verified 2011-02

CONDITIONS: Immobility and Weakness Associated With Long Intensive Care Unit Stays
Keywords: ICU LOS; Progressive Mobility; Deconditioning

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 4 months of observation: CVICU

SUMMARY:
The current study is proposed to assess the frequency and type of progressive mobility procedures currently performed in the CVICU The study will evaluate the type and frequency of progressive mobility orders, whether or not progressive mobility steps are being taken by the nursing teams, define what steps patients are receiving, and record time to first weight bearing. Other outcome measures will be the days of required mechanical ventilation, and current ICU length of stay and cost to treat.

DETAILED DESCRIPTION:
This will be a descriptive 4 month study of standard care practice. Patients who meet the inclusion / exclusion criteria for study will be enrolled (Waiver of informed consent is requested) and followed for a maximum of 28 days. The type and frequency of progressive mobility orders, whether or not progressive mobility steps are being taken by the nursing teams, define what steps patients are receiving, and record time to first weight bearing will be recorded. Weight bearing will be defined as standing for at least 1 minute. ICU LOS, Ventilator Days will be assessed at ICU discharge for study patients. Barriers to PM procedures will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Patient is ≥ 18 years old.
* Patient has been admitted to the ICU for less than 3 days prior to study enrollment
* Patients require mechanical ventilation for >48 hours

Exclusion Criteria:

* Mobilization is contraindicated by Patient's condition. Such as hip fractures or other injury that would impede standing posture.
* Patient weighs less than 70 pounds or more than 440 pounds
* Mobilization is contraindicated by patient's condition or physician's orders exist that prevent the patient from participating in the mobility protocol.
* Patient was unable to walk or stand without assistance prior to ICU admission.
* Patient was cognitively unable to follow verbal commands prior to ICU admission.
* Patients current diagnosis includes acute stroke with neurologic impairment
* Patient's current diagnosis includes drug overdose.
* Patient has "Do not resuscitate" orders and/or is at an end stage terminal disease state.
* Patient requires a specialty bed or mattress.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of patients admitted to the CV-Intensive Care Unit.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2010-07; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
First OOB | Days
  The ICU day that the patient is able to stand for at least 1 minute will be assessed.

SECONDARY OUTCOMES:
ICU LOS | Days
  Length of stay will be measured
Type and Frequency of PM orders | Daily
  The type and frequency of Progressive mobility orders will be assessed

CONTACTS AND LOCATIONS:
Overall Officials: Leslie Culpepper, MSN, RN, Principal Investigator — The Medical Cneter of Central Georgia
Locations (1):
- Medical College of Central Georgia, Macon, Georgia, United States